CLINICAL TRIAL: NCT01883492
Title: A Prospective Multi-center Randomized Study on Total Hip Replacement With E1
Brief Title: A Prospective Multi-center Study on Total Hip Arthroplasty With E1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment of the subject could not reach statistically required number.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INT.CR.GH2
Record Dates: First submitted 2013-01-31; First posted 2013-06-21 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Hip Osteoarthritis
Keywords: Only Female; Age between 20 - 75 at the time of operation
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BIOLOX delta head (Experimental): Uncemented Femoral Stem is inserted into femoral medullary canal. Uncemented Acetabular Cup is inserted into acetabular cavity with or without fixation screw(s).
  Acetabular Liner, which is made of E1 highly crosslinked polyethylene, is fitted into Acetabular cup.
  Biolox delta head is inserted onto the taper of the Femoral stem, and is articulating against Acetabular Liner made of E1.
  Interventions: Device: Femoral Stem; Device: Acetabular Cup; Device: Acetabular Liner
- CoCr head (Active Comparator): Uncemented Femoral Stem is inserted into femoral medullary canal. Uncemented Acetabular Cup is inserted into acetabular cavity with or without fixation screw(s).
  Acetabular Liner, which is made of E1 highly crosslinked polyethylene, is fitted into Acetabular cup.
  CoCr head is inserted onto the taper of the Femoral stem, and is articulating against Acetabular Liner made of E1.
  Interventions: Device: Femoral Stem; Device: Acetabular Cup; Device: Acetabular Liner

INTERVENTIONS:
Device: Femoral Stem — JMDN classification/Class III device
  Other Names: Taperloc Complete; Taperloc Microplasty Complete; Taperloc Complete XR123; Taperloc Microplasty Complete XR123
Device: Acetabular Cup — JMDN classification: Class III device
  Other Names: Ringloc Acetabular Cup; Regenerex Ringloc+ Acetabular Cup
Device: Acetabular Liner — JMDN classification: Class III device
  Other Names: E1 Ringloc Liner

SUMMARY:
The primary objectives of this clinical study include:

* Evaluate E1 Wear including early bedding-in process, clinical outcomes on patients who received Total Hip Arthroplasty with E1
* Compare E1 wear used with CoCr and Biolox Delta heads

DETAILED DESCRIPTION:
This study is designed as PROSPECTIVE, RANDOMIZED, MULTI-CENTER Study to compare two different materials (CoCr and Delta ceramic) articulating against E1 Highly Crosslinked polyethylene in Hip Replacement.

Patient population is 160 (80 each). Follow-up period is 10 year postoperatively. E1 liners with thickness of 4.8mm at 45 degrees position (load bearing direction) will be used in all cases.

Randomization will occur via random number generator by 4 blocks randomization.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis
* Age between 20 - 75 at the time of operation
* Patients with limited co-morbidity -ASA I-III
* Patients must be able to understand instructions and be willing to return for follow up

Exclusion Criteria:

* In accordance with approved Absolute and Relative Contraindications for use in participating countries for E1 liner and Delta Ceramic and CoCr femoral head hip system System.

Absolute contraindications include: infection, sepsis, and osteomyelitis.

Relative contraindications include:

1. uncooperative patient or patient with neurologic disorders who are incapable of following directions,
2. osteoporosis,
3. metabolic disorders which may impair bone formation,
4. osteomalacia,
5. distant foci of infections which may spread to the implant site,
6. rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram, and
7. vascular insufficiency, muscular atrophy, or neuromuscular disease.
8. pregnancy

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hirotsugu Ohashi, M.D., Ph.D., Principal Investigator — Saiseikai Nakatsu Hospital; Arihiko Kanaji, M.D., Ph.D., Principal Investigator — Keio University; Katsufumi Uchiyama, M.D., Ph.D., Principal Investigator — Kitasato University School of Medicine; Hironori Kaneko, M.D., Ph.D., Principal Investigator — Kitasato University Kitasato Institute Hospital; Koichi Kinoshita, M.D., Ph.D., Principal Investigator — Fukuoka University School of Medicine
Locations (5):
- Japan (5):
  - Fukuoka University School of Medicine, Fukuoka, Fukuoka
  - Kitasato University School of Medicine, Sagamihara, Kanagawa
  - Saiseikai Nakatsu Hospital, Osaka
  - Kitasato University Kitasato Institute Hospital, Tokyo
  - Keio University School of Medicine, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BIOLOX Delta Head: Uncemented Femoral Stem is inserted into femoral medullary canal. Uncemented Acetabular Cup is inserted into acetabular cavity with or without fixation screw(s).
  Acetabular Liner, which is made of E1 highly crosslinked polyethylene, is fitted into Acetabular cup.
  Biolox delta head is inserted onto the taper of the Femoral stem, and is articulating against Acetabular Liner made of E1.
  Femoral Stem: JMDN classification/Class III device
  Acetabular Cup: JMDN classification: Class III device
  Acetabular Liner: JMDN classification: Class III device
- CoCr Head: Uncemented Femoral Stem is inserted into femoral medullary canal. Uncemented Acetabular Cup is inserted into acetabular cavity with or without fixation screw(s).
  Acetabular Liner, which is made of E1 highly crosslinked polyethylene, is fitted into Acetabular cup.
  CoCr head is inserted onto the taper of the Femoral stem, and is articulating against Acetabular Liner made of E1.
  Femoral Stem: JMDN classification/Class III device
  Acetabular Cup: JMDN classification: Class III device
  Acetabular Liner: JMDN classification: Class III device
Period: Overall Study
Arm/Group | BIOLOX Delta Head | CoCr Head
Started | 75 | 78
Completed | 62 | 67
Not Completed | 13 | 11
Not completed — Lost to Follow-up | 3 | 4
Not completed — Surgery on contra-lateral hip | 0 | 1
Not completed — Poor X-ray quality | 7 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — inappropriate implant used | 1 | 1
Not completed — bone anatomy did not meet study criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIOLOX Delta Head | CoCr Head | Total
Number analyzed (Participants) | 62 | 67 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.90 (7.16) | 61.94 (7.26) | 61.92 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 67 | 129
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 62 | 67 | 129
Harris Hip Score [Mean (Standard Deviation); unit: score on scale] — Harris Hip Score is Physician rating score to evaluate hip disabilities. Score domains are "pain", "function", "absence of deformity" and "range of hip motion".
  Minimum possible score is 0 and maximum possible score is 100. Higher score means better outcome.
  score on scale | 55.11 (11.65) | 52.63 (11.67) | 53.83 (11.68)
WOMAC osteoarthritis index [Mean (Standard Deviation); unit: score on scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is used in evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items.
  The scores for each subscale are summed up, with a possible score range of 0-20 for "Pain", 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a The total WOMAC score ranged from 0 to 96.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
  score on scale | 40.75 (17.09) | 41.24 (15.29) | 41.00 (16.13)
UCLA Activity Score [Mean (Standard Deviation); unit: score on scale] — University of California, Los Angeles (UCLA) activity score is questionnaire to assess intensity of patients' activity.
  The score ranges from 1 to 10 (1 point increment), higher score means higher activity level.
  score on scale | 2.95 (0.95) | 3.28 (1.10) | 3.12 (1.04)

OUTCOME MEASURES:

1. Primary Outcome: Polyethylene Wear Between Immediate Postoperative and 2 Year Postoperative Period
Description: Vector wear, which is defined as movement (difference of femoral prosthetic head positions) between immediate postoperative and 2 years postoperative periods. There is no lower and upper limit, actual measured results. The outcome can be negative value.
Time Frame: Immediate postoperative and 2 year postoperatively
Population: Participants, whose x-ray taken at 2 year follow-up visit being available.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 57 | 63
millimeter | 0.42 (1.08) | 0.15 (0.70)

2. Secondary Outcome: Harris Hip Score at 6 Month Follow-up Visit
Description: Harris Hip Score is Physician rating score to evaluate hip disabilities. Score domains are "pain", "function", "absence of deformity" and "range of hip motion".
  Minimum possible score is 0 and maximum possible score is 100. Higher score means better outcome.
Time Frame: 6 month postoperative
Population: 1 patient in BIOLOX delta head group and 13 patients in CoCr head group missed collecting Harris Hip Score at 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 61 | 54
score on a scale | 92.67 (8.05) | 92.61 (7.92)

3. Secondary Outcome: Harris Hip Score at 1 Year Follow-up Visit
Description: as for outcome 2
Time Frame: 1 year postoperative
Population: 1 patient in BIOLOX delta head group and 6 patients in CoCr head group missed collecting Harris Hip Score at 1 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 61 | 61
score on a scale | 95.23 (6.10) | 94.52 (6.76)

4. Secondary Outcome: Harris Hip Score at 2 Year Follow-up Visit
Description: as for outcome 2
Time Frame: 2 year postoperative
Population: 3 patients in BIOLOX delta head group and 9 patients in CoCr head group missed collecting Harris Hip Score at 2 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 59 | 58
score on a scale | 96.15 (5.44) | 96.28 (5.69)

5. Secondary Outcome: Harris Hip Score at 3 Year Follow-up Visit
Description: as for outcome 2
Time Frame: 3 year postoperative
Population: 12 patients in BIOLOX delta head group and 12 patients in CoCr head group missed collecting Harris Hip Score at 3 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 50 | 55
score on a scale | 96.30 (4.56) | 96.82 (6.03)

6. Secondary Outcome: WOMAC Osteoarthritis Index at 6 Month Follow-up Visit
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is used in evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items.
  The scores for each subscale are summed up, with a possible score range of 0-20 for "Pain", 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a The total WOMAC score ranged from 0 to 96.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: 6 month postoperative
Population: 6 patients in BIOLOX delta head group and 11 patients in CoCr head group missed colleting WOMAC questionnaire at 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 56 | 56
score on a scale | 9.27 (9.75) | 10.43 (9.62)

7. Secondary Outcome: WOMAC Osteoarthritis Index at 1 Year Follow-up Visit
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is used in evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items.
  The scores for each subscale are summed up, with a possible score range of 0-20 for "Pain", 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a The total WOMAC score ranged from 0 to 96.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: 1 year postoperative
Population: 6 patients in BIOLOX delta head group and 13 patients in CoCr head group missed colleting WOMAC questionnaire at 1 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 56 | 54
score on a scale | 9.86 (13.52) | 9.57 (9.23)

8. Secondary Outcome: WOMAC Osteoarthritis Index at 2 Year Follow-up Visit
Description: as for outcome 7
Time Frame: 2 year postoperative
Population: 9 patients in BIOLOX delta head group and 16 patients in CoCr head group missed colleting WOMAC questionnaire at 2 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 53 | 51
score on a scale | 7.85 (8.88) | 7.80 (10.32)

9. Secondary Outcome: WOMAC Osteoarthritis Index at 3 Year Follow-up Visit
Description: as for outcome 7
Time Frame: 3 year postoperative
Population: 14 patients in BIOLOX delta head group and 17 patients in CoCr head group missed colleting WOMAC questionnaire at 3 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 48 | 50
score on a scale | 8.29 (9.31) | 6.84 (8.00)

10. Secondary Outcome: UCLA Activity Score at 6 Month Follow-up Visit
Description: University of California, Los Angeles (UCLA) activity score is questionnaire to assess intensity of patients' activity.
  The score ranges from 1 to 10 (1 point increment), higher score means higher activity level.
Time Frame: 6 month postoperative
Population: 4 patients in BIOLOX delta head group and 12 patients in CoCr head group missed colleting UCLA Activity score at 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 58 | 55
score on a scale | 5.19 (1.42) | 4.75 (1.28)

11. Secondary Outcome: UCLA Activity Score at 1 Year Follow-up Visit
Description: as for outcome 10
Time Frame: 1 year postoperative
Population: 2 patients in BIOLOX delta head group and 8 patients in CoCr head group missed colleting UCLA Activity score at 1 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 60 | 59
score on a scale | 5.45 (1.52) | 5.03 (1.27)

12. Secondary Outcome: UCLA Activity Score at 2 Year Follow-up Visit
Description: as for outcome 10
Time Frame: 2 year postoperative
Population: 3 patients in BIOLOX delta head group and 9 patients in CoCr head group missed colleting UCLA Activity score at 2 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 59 | 58
score on a scale | 5.53 (1.38) | 5.31 (1.30)

13. Secondary Outcome: UCLA Activity Score at 3 Year Follow-up Visit
Description: as for outcome 10
Time Frame: 3 year postoperative
Population: 12 patients in BIOLOX delta head group and 11 patients in CoCr head group missed colleting UCLA Activity score at 3 year visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BIOLOX Delta Head | CoCr Head
Number analyzed (Participants) | 50 | 56
score on a scale | 5.42 (1.49) | 5.43 (1.36)

ADVERSE EVENTS:
Time Frame: 3 year after surgery
Arm/Group | BIOLOX Delta Head | CoCr Head
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/67
Other Adverse Events (participants affected / at risk) | 2/62 | 1/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOLOX Delta Head (N=62) | CoCr Head (N=67)
Intraoperative Trochanteric Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Surgical Procedure related intraoperative fracture of Trochanter of Femur.
Femoral Nerve Palsy (Nervous system disorders) | 1 (1) | 0 (0) — Surgical Procedure related femoral nerve palsy. Symptom was disappeared although no specific treatment was conducted.
Inappropriate femoral stem position (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Intraoperative stem insertion to prepared femoral canal was not optimal, so it was revised two weeks after primary surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-02-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT01883492/Prot_SAP_000.pdf